CLINICAL TRIAL: NCT00930202
Title: Open Label Study of the Safety and Efficacy of Conivaptan (Vaprisol®) to Raise Serum Sodium Levels in Patients With Severe Traumatic Brain Injury
Brief Title: Study of the Safety and Efficacy of Conivaptan (Vaprisol®) to Raise Serum Sodium Levels in Patients With Severe Traumatic Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Miriam Treggiari, Associate Professor of Anesthesiology & Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35774-A
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Severe Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Conivaptan; Vaprisol; Sodium
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — conivaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conivaptan (Vaprisol) (Experimental): Conivaptan (Vaprisol) will be administered in a single dose of 20 mg, mixed with 100 mL of 5% dextrose in water, and delivered over 30 minutes.
  Interventions: Drug: Conivaptan (Vaprisol)
- Standard Care (No Intervention): No intervention

INTERVENTIONS:
Drug: Conivaptan (Vaprisol) — Conivaptan (Vaprisol) will be administered in a single dose of 20 mg, mixed with 100 mL of 5% dextrose in water, and delivered over 30 minutes.
  Arms: Conivaptan (Vaprisol)

SUMMARY:
The investigators plan to utilize conivaptan (Vaprisol) to promote isolated water loss, in combination with normal (physiologic) fluid replacement to maintain a normal blood volume status, in patients with severe TBI. The goal of this therapy is to raise blood sodium in a controlled fashion in subjects with severe TBI, and reduce the use of hypertonic saline infusion. We hypothesize that this therapy will maintain a stable state of high blood sodium, while decreasing the overall sodium load needed to achieve these goals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* Initial diagnosis of an isolated, severe traumatic brain injury (Glasgow Coma Score of 8 or less upon initial evaluation)
* Cerebral edema with a head CT and Marshall classification of diffuse injury type II, III, or IV.
* Primary care team orders to raise blood sodium by 10 mEq/L from baseline.
* Placement of an intraparenchymal fiberoptic monitor to monitor intracranial pressure (ICP).

Exclusion Criteria:

* Age < 18 years
* Signs of hypovolemia including systolic BP < 90 mmHg
* Signs of liver disease including jaundice and ascites

  * AST > 35 units/L
  * ALT > 35 units/L
* Signs of renal disease including history of dialysis

  * Serum creatinine > 1.5 mg/dL
  * BUN > 20 mg/dL range
* Baseline serum sodium >/= 145 mEq/L
* Pregnant or lactating females
* Concomitant use of digoxin, ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, simvastatin and lovastatin
* Presentation to the tertiary care hospital > 24 hours post-injury
* Multi-system traumatic injuries
* Diabetes Insipidus
* Anticipation of diagnosis compatible with brain death, or no expectation of survival with 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of events of excessive rate of increase in sodium levels (>1 mEq/hr). | Every 4 hours

SECONDARY OUTCOMES:
Safety profile: number of events of increased serum sodium levels above the intended target range, and any adverse events occurring during the study period. | Hospital Stay
Sodium load: Sodium load is defined as the cumulative amount of sodium administered by enteral and parenteral routes from the time of randomization to 48 hours post-randomization | Until 48 hours post randomization
Serum sodium stability: a. Stable state of hypernatremia b. Sodium variability c. Time to achievement of target sodium levels after randomization | Until 48 hours post randomization
Fluid balance | Until 48 hours post randomization
Cerebral edema: a. Mean ICP in the first 48 hours after randomization b. Reduction of cerebral edema | Until 48 hours post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States